CLINICAL TRIAL: NCT06669533
Title: Misoprostol to Optimizing Prevention of Cancer of the Cervix: A Double-Blind Randomized Controlled Trial
Brief Title: Use Misoprostol to Optimize Prevention of Cervical Cancer
Acronym: MISOPCx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Cameroon Baptist Convention Health Core (Unknown)
Responsible Party: Principal Investigator, Warner Huh, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB-30012879; 1R01CA279021 (NIH)
Record Dates: First submitted 2024-10-18; First posted 2024-11-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-07

CONDITIONS: Cervical Cancers
Keywords: cervical cancers
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Misoprostol

STUDY DESIGN:
Masking Description: The PIs, nurses who will be providing the drugs, and study participants will be blinded in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Non-pregnant women (Experimental): Non-pregnant women will either receive 600 mcg misoprostol (3 tablets) or identical placebo 3 (tablets) administered vaginally 2-3 hours and 4-6 hours prior to visual inspection with acetic acid (VIA).
  Interventions: Drug: Placebo; Drug: Misoprostol

INTERVENTIONS:
Drug: Placebo — Participants will receive placebo (3 tablets) administered vaginally 2-3 hours and 4-6 hours prior to visual inspection with acetic acid (VIA).
Drug: Misoprostol — Participants will receive 600 mcg misoprostol (3 tablets) administered vaginally 2-3 hours and 4-6 hours prior to visual inspection with acetic acid (VIA).

SUMMARY:
This is a double-blind randomized controlled trial of 420 non-pregnant women undergoing cancer screening by visual inspection with acetic acid (VIA) who have Type 3 transformation zone (TZ) and randomized to receive either Misoprostol or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 3 TZ confirmed on exam prior to randomization
* Age 25 years or older

Exclusion Criteria:

* With Type 1 or 2 TZ prior to randomization
* Currently pregnant
* History of hysterectomy
* Any cancerous lesions
* Active cervicitis

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Non-pregnant women
Enrollment: 420 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-11-04 (Estimated); Study Completion 2027-11-04 (Estimated)

PRIMARY OUTCOMES:
Conversion rate from Type 3 transformation zone (TZ) to Types 1 or 2 | Approximately 2-3 hours and approximately 4-6 hours since drug administration
  The rate of participants with successful transformation from Type 3 (TZ) to Type 1 or 2 (TZ) will be calculated. It is the number of participants who successfully transformed from Type 3 TZ to Type 1 or 2 TZ, divided by the total number of participants in the entire randomized cohort.

SECONDARY OUTCOMES:
Comparison of the rate of patients converted from Type 3 TZ to Type 1 or 2 TZ between 2-3 hours and 4-6 hours | Approximately 2-3 hours vs approximately 4-6 hours
  The rate of transformation from Type 3 transformation zone (TZ) to Type 1 or 2 TZ between 2-3 hours and 4-6 hours after administering misoprostol will be compared. The rate is calculated as the number of successful transformations within each time period (2-3 hours or 4-6 hours) divided by the total cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Warner K Huh, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Cameroon Baptist Convention Health Core, EtougEbe Baptist Hospital Yaoundé, Yaoundé, Center Region, Cameroon

IPD SHARING:
Plan to Share IPD: Undecided